CLINICAL TRIAL: NCT00387998
Title: Randomized Trial of a Primer to Help Patients Understand Risk
Brief Title: Health Education in Improving the Understanding of Medical Information
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: CDR0000510867; R18CA091052 (NIH); DMS-15144; NCT00380432 (obsolete NCT alias)
Record Dates: First submitted 2006-10-12; First posted 2006-10-13 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2008-01

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Risk primer (Experimental): Booklet written by investigators "know your chances"
  Interventions: Other: Risk primer
- Control booklet (Active Comparator): AHRQ staying healthy booklet
  Interventions: Other: AHRQ staying healthy booklet

INTERVENTIONS:
Other: AHRQ staying healthy booklet — educational booklet about prevention
  Other Names: AHRQ guide to staying healthy
  Arms: Control booklet
Other: Risk primer — Know your chances booklet
  Other Names: Know your chances
  Arms: Risk primer

SUMMARY:
RATIONALE: Understanding the risk of disease and prevention and screening activities to lower disease risk may help individuals make informed medical decisions.

PURPOSE: This randomized clinical trial is studying how well health education materials help participants understand medical information.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare medical data interpretation skills in participants of low or high socioeconomic status who receive a general education primer (entitled "Know Your Chances: Understanding Health Statistics") vs a health education booklet (entitled "The Pocket Guide to Good Heath for Adults").

OUTLINE: This is a randomized, controlled study. Participants are stratified according to socioeconomic status (low vs high). Participants are randomized to 1 of 2 intervention arms.

* Arm I (control): Participants receive a health education booklet entitled "The Pocket Guide to Good Health for Adults," published by the Agency for Health Care Research and Quality, which contains general information about disease risk and reducing risk by following recommended prevention or screening activities.
* Arm II (primer): Participants receive a general education primer entitled "Know your chances: Understanding health statistics," which teaches how to understand disease risk and the benefits and risks of intervention.

Within 2 weeks after receiving the education material, participants in both arms complete a survey, including a medical data interpretation test, STAT-interest, STAT-confidence, and user ratings of the education materials.

PROJECTED ACCRUAL: A total of 555 participants were accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * High socioeconomic status

    * Attended Dartmouth Community Medical School in the past
  * Low socioeconomic status

    * Veteran or family member enrolled in a Veteran Affairs clinic

PATIENT CHARACTERISTICS:

* English speaking
* No more than 1 participant per household

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 35 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 555 (Actual)
Dates: Start 2004-10; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Ability to interpret medical statistics as measured by a medical data interpretation test | 2 weeks
  medical data interpretation skills

SECONDARY OUTCOMES:
Interest in interpreting medical statistics, as measured by STAT-interest | 2 weeks
  STAT-interest measure
Confidence in interpreting medical statistics, measured by STAT-confidence | 2 weeks
  STAT-confidence
User ratings of materials | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Steven Woloshin, MD, MS, Principal Investigator — White River Junction Veterans Affairs Medical Center; Lisa Schwartz, MD, MS, Principal Investigator — White River Junction Veterans Affairs Medical Center

REFERENCES:
- [Derived] Woloshin S, Schwartz LM, Welch HG. The effectiveness of a primer to help people understand risk: two randomized trials in distinct populations. Ann Intern Med. 2007 Feb 20;146(4):256-65. doi: 10.7326/0003-4819-146-4-200702200-00004. PMID 17310049